CLINICAL TRIAL: NCT00442156
Title: The Course of Response to Focal Photocoagulation for Diabetic Macular Edema
Brief Title: The Course of Response to Focal Photocoagulation for DME
Acronym: Laser Resp
Status: Completed | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Roy W. Beck, M.D., Ph.D., Director, Jaeb Center for Health Research (DRCR.net)
Other Study IDs: NEI-131; U10EY018817-03 (NIH); U10EY014229-07 (NIH); U10EY014231-09 (NIH)
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema
Keywords: Laser photocoagulation
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Lasers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Laser: People with diabetic macular edema involving the center of the macula (OCT central subfield thickness >250 microns), who were already intended to receive focal photocoagulation
  Interventions: Procedure: Laser photocoagulation

INTERVENTIONS:
Procedure: Laser photocoagulation — modified ETDRS focal photocoagulation generally completed in a single sitting on the day of enrollment, but if little or no improvement, may be repeated at 16 weeks
  Other Names: Laser

SUMMARY:
The study objective is to determine the course of changes in OCT measured macular thickness and visual acuity following a single session of focal photocoagulation for center-involved DME. The response will be evaluated separately in eyes with and without prior focal photocoagulation for DME. The purpose is to determine the proportion of eyes that continue to improve at least 5 letters in visual acuity or at least 10% in central retinal thickness after a session of focal photocoagulation. In addition, the study will explore whether any baseline factors can be identified that are predictive of the response.

All subjects will have follow-up visits 8 weeks and 16 weeks post treatment. At the 16-week visit, study eyes are evaluated for change in retinal thickness and visual acuity from baseline.

* Treatment is to be deferred and follow up continued if visual acuity letter score has improved by >5 or OCT central subfield thickness has decreased by >10% compared with baseline.
* If visual acuity letter score has not improved by at least 5 and OCT central subfield thickness has not decreased by at least 10%, then the eye is classified as 'not improved' and the investigator may provide additional treatment. Follow up ends for eyes that receive additional treatment at this visit. However, if the investigator and participant elect to defer additional treatment (even if deferral criteria are not met), then follow up will continue until the study eye receives additional treatment for DME.
* Eyes continuing in follow up have visits every 8 weeks (+1week) as long as there has been continued improvement in visual acuity (letter score improved >5 ) or retinal thickness (central subfield thickness decreased by >10%) compared with the visit 16 weeks earlier. The longest follow-up time will be 48 weeks.

By providing information on the length of time during which clinically meaningful improvement occurs following focal photocoagulation, clinicians will be better able to determine when further photocoagulation or other treatments should be considered for persistent DME. Depending on the results of this study, a future randomized clinical trial will be considered comparing the more aggressive retreatment photocoagulation regimen currently serving as the standard DRCR Network approach to focal photocoagulation for macular edema with the less aggressive regimen evaluated in this protocol.

DETAILED DESCRIPTION:
Focal photocoagulation is the only treatment that has been demonstrated to be beneficial for diabetic macular edema. In the ETDRS, focal photocoagulation of eyes with macular edema reduced the risk of moderate visual loss (decrease of 15 or more letters) by approximately 50% (from 24% to 12%, three years after initiation of treatment). For eyes with center-involved DME and visual acuity worse than 20/40 that were treated with focal photocoagulation, the 15-letter improvement rate at 1 year was 11% and at 3 years was 16%.

In the ETDRS, focal photocoagulation treatment for diabetic macular edema involved direct treatment to discrete lesions between 500 microns and 3000 microns from the center of the macula that were thought to be causing retinal thickening or hard exudates with or without "grid" treatment to other macular areas of retinal thickening or non-perfusion. The lesions treated directly included microaneurysms, identified on fluorescein angiography, that either filled or leaked, intraretinal microvascular abnormalities (IRMA), or pruned capillaries that leaked fluorescein. Grid treatment was applied in the ETDRS to areas of thickened retina that showed diffuse fluorescein leakage or areas of non-perfusion identified as capillary dropout on fluorescein angiography. Areas of non-perfusion in the macula could be treated with grid at the discretion of the treating ophthalmologist. Areas that had both discrete lesions and diffuse leakage or capillary dropout would receive a combination of direct and grid treatment. Re-treatment was applied at four month intervals if clinically significant macular edema persisted, one or more treatable lesions were identified, and the investigator believed these lesions were responsible for the edema. The median number of focal laser treatments applied in the ETDRS was 3.8.

The mechanism of action of focal photocoagulation is not fully understood; however, it is clear that the retinal pigment epithelium (RPE) absorbs the majority of the laser energy and thermal injury occurs at the level of the RPE. Studies have shown that photocoagulation can eventually result in retinal and apparent RPE atrophy 200-300% larger than the original laser spot size. These areas of expanded atrophy can lead to loss of central vision, central scotomata, and decreased color vision. Consequently, many retinal specialists today tend to treat with lighter, less intense laser burns than originally specified in the ETDRS.

In addition to the concern regarding the spread of intense laser burns, there are a number of other reasons that retinal specialists today have modified the treatment procedures originally specified in the ETDRS protocol. These reasons include the advent of new lasers and the clinical observation that different techniques, such as focal photocoagulation with lighter burns or grid treatment alone, may be similar in beneficial effect as the original ETDRS treatment protocol. A modified ETDRS focal photocoagulation protocol adapted from the original ETDRS approach, has been adopted as the standard laser technique for DME used in DRCRnet studies.

There are limited data on the course of visual acuity and central retinal thickness after a single focal photocoagulation session for DME. In prior DRCRnet DME treatment protocols that included a laser arm, according to the re-treatment protocol eyes received a second focal photocoagulation session at 3.5- 4 months (which was the first follow-up visit) unless there was substantial improvement defined as at least a 50% decrease in retinal thickening of the central subfield measurement on OCT. As a result, it is unknown what proportion of eyes with lesser degrees of improvement would have continued to improve and the time course for further improvement following the initial photocoagulation session given additional time. In one study conducted by DRCRnet of eyes that had not been previously treated for DME, among 113 eyes in the modified ETDRS laser treatment group with baseline OCT central subfield >250 microns, a 50% or more reduction in OCT central subfield thickening was present at 3.5 months in only 28 (25%). The table below categorizes the 85 eyes that did not meet this measure of improvement at 3.5 months with regard to improvement in visual acuity of at least 5 letters and/or reduction in central subfield thickness of at least 10%. The 5 letter reduction was selected based on the 95% confidence interval for change determined in a study that evaluated the validity and reliability of the electronic ETDRS visual acuity testing procedure that is used in DRCRnet protocols. The 10% threshold was selected based on the DRCRnet OCT reproducibility study which found that a 10% change in central subfield thickness was likely to be real. Forty-seven (42%) eyes that met the protocol requirement for repeat photocoagulation at the first follow-up visit had an improvement in either visual acuity (of at least 5 letters), central subfield (of at least a 10% reduction), or both at this follow-up visit.

Other DRCRnet protocols provide data on the course following a single photocoagulation session through 4 months of follow up. In a pilot study designed to evaluate peribulbar corticosteroids for mild DME (OCT central subfield thickness = 250 microns and visual acuity 20/40 or better at baseline), modified ETDRS focal photocoagulation was the treatment given to the control group. Follow-up visits occurred after 1, 2, and 4 months before the eye was eligible to be retreated. Twenty-one of the 37 eyes in the laser group had not been previously treated with focal photocoagulation for DME and 17 eyes had been previously treated with focal photocoagulation. A 50% or more reduction in OCT central subfield thickening occurred in 11 (30%) of the 37 eyes at 17 weeks. Fourteen (38%) eyes that would have met the criteria for re-treatment had an improvement in either visual acuity (of at least 5 letters), central subfield (of at least 10%), or both at 17 weeks.

In another pilot study evaluating intravitreal bevacizumab for DME (OCT central subfield thickness = 275 microns and visual acuity 20/32 or worse at baseline), modified ETDRS focal photocoagulation was the treatment given to the control group. Follow-up visits occurred after 3, 6, 9, and 12 weeks before the eye was eligible to be retreated. There were 7 eyes in the laser group that had not been previously treated with focal photocoagulation for DME and 12 eyes that had been previously treated with focal photocoagulation. Among these 19 eyes, a 50% or more reduction in OCT central subfield thickening occurred in 3 (16%) at 12 weeks. Ten (53%) eyes that would have met criteria for re-treatment had an improvement in either visual acuity (of at least 5 letters), central subfield (of at least 10%), or both at 12 weeks.

The data from these three protocols indicate that a substantial number of eyes receiving focal photocoagulation (either an initial course or repeat application) will show improvement in central retinal thickness after 3-4 months that is at least 10% but is less than 50% of the baseline thickening. It is for these eyes that further knowledge of the course of retinal thickening and visual acuity without additional interventions is needed to assess whether the present requirements for re-treatment are more aggressive than they need to be.

ELIGIBILITY:
Inclusion Criteria

To be eligible, the following inclusion criteria must be met:

* Age >= 18 years
* Diagnosis of diabetes mellitus (type 1 or type 2.
* At least one eye meets the study eye criteria.
* Able and willing to provide informed consent.

The subject must have one eye meeting all of the inclusion criteria and none of the exclusion criteria listed below. If both eyes are eligible, the study eye is selected by the investigator and subject.

* Best corrected E-ETDRS visual acuity letter score >= 24 (i.e., 20/320 or better) within 8 days of enrollment.
* On clinical exam, definite retinal thickening due to diabetic macular edema involving the center of the macula.
* OCT central subfield >=250 microns within 8 days of enrollment.
* Media clarity, pupillary dilation, and subject cooperation sufficient for adequate OCT.
* Investigator believes that focal photocoagulation is the most appropriate treatment for the DME.
* Study Eye Exclusion Criteria

Exclusion Criteria

A subject is not eligible if any of the following exclusion criteria are present:

* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
* Blood pressure > 180/110 (systolic above 180 OR diastolic above 110).
* Participation in an investigational trial within 30 days of enrollment that involved treatment with any drug that has not received regulatory approval at the time of study entry.
* Subject is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the next 6 months.

The following exclusions apply to the study eye only (i.e., they may be present for the nonstudy eye):

* Macular edema is considered to be due to a cause other than diabetic macular edema.
* An ocular condition is present such that, in the opinion of the investigator, visual acuity loss would not improve from resolution of macular edema (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, significant macular ischemia, nonretinal condition).
* An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.).
* Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal).
* History of treatment for DME at any time in the past 4 months (such as focal/grid macular photocoagulation, intravitreal or peribulbar corticosteroids, anti-VEGF drugs, or any other treatment).
* History of panretinal (scatter) photocoagulation (PRP) within 4 months prior to enrollment or anticipated to be performed within next 6 months.
* History of major ocular surgery (including vitrectomy, cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 4 months or anticipated within the next 6 months.
* History of YAG capsulotomy performed within 2 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetics within the United States who are at least 18 years old and have DME treatable with laser photocoagulation.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
OCT-measured retinal thickness and visual acuity | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Browning, M.D., Study Chair — Charlotte Eye, Ear, Nose and Throat Assoc., PA
Locations (32):
- United States (32):
  - Southern California Desert Retina Consultants, MC, Palm Springs, California
  - Retina Vitreous Consultants, Fort Lauderdale, Florida
  - Retina Consultants of Southwest Florida, Fort Myers, Florida
  - Central Florida Retina Institute, Lakeland, Florida
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Retina Associates of Hawaii, Inc., Honolulu, Hawaii
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - American Eye Institute, New Albany, Indiana
  - Retina and Vitreous Associates of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Maine Vitreoretinal Consultants, Bangor, Maine
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Southern New England Retina Associates, Attleboro, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - Associated Retina Consultants, Williamsburg, Michigan
  - Delaware Valley Retina Associates, Lawrenceville, New Jersey
  - University of Rochester, Rochester, New York
  - Retina-Vitreous Surgeons of Central New York, PC, Syracuse, New York
  - University of North Carolina, Dept. of Ophthalmology, Chapel Hill, North Carolina
  - Charlotte Eye, Ear, Nose and Throat Assoc., PA, Charlotte, North Carolina
  - Retina Associates of Cleveland, Inc., Beachwood, Ohio
  - Casey Eye Institute, Portland, Oregon
  - Palmetto Retina Center, Columbia, South Carolina
  - Carolina Retina Center, Columbia, South Carolina
  - Retina Research Center, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Charles A. Garcia, PA & Associates, Houston, Texas
  - Retina and Vitreous of Texas, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - University of Wisconsin-Madison, Dept. of Ophthalmology, Madison, Wisconsin

REFERENCES:
- [Result] Diabetic Retinopathy Clinical Research Network. The course of response to focal/grid photocoagulation for diabetic macular edema. Retina. 2009 Nov-Dec;29(10):1436-43. doi: 10.1097/IAE.0b013e3181bcef6b. PMID 19898182